CLINICAL TRIAL: NCT04214119
Title: EsophaCap for the Detection of Early Esophageal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00072332; R01DK118250 (NIH)
Record Dates: First submitted 2019-12-26; First posted 2020-01-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Barrett Esophagus; Esophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Esophageal and gastric brush cells.
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (4):
- Control: Patients age 18 or greater who have undergone esophagogastroduodenoscopy and does not have a diagnosis of Barrett's esophagus or esophageal/gastric malignancy.
- Barrett's esophagus: Patients age 18 or greater who have undergone esophagogastroduodenoscopy and diagnosed with Barrett's esophagus via pathology.
- Esophageal carcinoma: Patients age 18 or greater who have diagnosis of primary esophageal carcinoma.
- Gastric cancer: Patients age 18 or greater who have diagnosis of primary esophageal cancer.

SUMMARY:
This study is to identify potential biomarkers for the early detection of Barrett's Esophagus, esophageal carcinoma (both adenocarcinoma and squamous cell carcinoma), and gastric cancer via sponge cytology.

DETAILED DESCRIPTION:
This study is to identify potential biomarkers for the early detection of Barrett's Esophagus, esophageal carcinoma (both adenocarcinoma and squamous cell carcinoma). Esophageal and gastric cytology will be collected via sponge capsule. Candidate genes will be tested with DNA isolated from these samples in order to identify optimal biomarkers to differentiate between Barrett's esophagus and esophageal/gastric cancer versus normal esophageal/gastric tissue.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing esophagogastroduodenoscopy at Johns Hopkins Hospital from 1/2016 to 12/2025
* Age greater than 18 years
* Patients must be able to swallow a capsule

Exclusion Criteria:

* Patients in either arm with extra-esophageal malignancies including head and neck and gastric cancer
* Patients who have undergone esophagectomy
* Patients who have undergone radiation to the chest
* Patients who are younger than 18
* Patients with esophageal stents
* Patients with esophageal strictures disabling passage of the capsule

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for clinically indicated upper endoscopy will be approached to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2016-01-12 (Actual); Primary Completion 2028-12-19 (Estimated); Study Completion 2028-12-19 (Estimated)

PRIMARY OUTCOMES:
Difference in methylation of gene markers to discriminate Barrett's esophagus from non-pathological esophageal squamous and gastric cardia tissue. | 1 day
  Using DNA methylation, we plan on identifying, from a pool of highly selected marker candidates, the best biomarkers that are aberrantly methylated in Barrett's esophagus versus control in order to differentiate between subjects who have Barrett's esophagus and those who do not have Barrett's esophagus. This is measure using methylation index and the calculated probability score from different methylation index values.
Difference in methylation of gene markers to discriminate esophageal carcinoma from non-pathological esophageal squamous and gastric cardia tissue. | 1 day
  Using DNA methylation, we plan on identifying, from a pool of highly selected marker candidates, the best biomarkers that are aberrantly methylated in esophageal cancer versus control in order to differentiate between subjects who have esophageal cancer and those who do not. This is measure using methylation index and the calculated probability score from different methylation index values.
Difference in methylation of gene markers to discriminate gastric cancer from non-pathological esophageal squamous and gastric cardia tissue. | 1 day
  Using DNA methylation, we plan on identifying, from a pool of highly selected marker candidates, the best biomarkers that are aberrantly methylated in gastric cancer versus control in order to differentiate between subjects who have gastric cancer and those who do not. This is measure using methylation index and the calculated probability score from different methylation index values.

SECONDARY OUTCOMES:
Sensitivity of candidate biomarker p16 | 1 day
  Sensitivity of each candidate biomarker will be calculated by measuring the area under receiver operating characteristic curve generated from methylation index data.
Sensitivity of candidate biomarker NELL1 | 1 day
  Sensitivity of each candidate biomarker will be calculated by measuring the area under receiver operating characteristic curve generated from methylation index data.
Sensitivity of candidate biomarker AKAP12 | 1 day
  Sensitivity of each candidate biomarker will be calculated by measuring the area under receiver operating characteristic curve generated from methylation index data.
Sensitivity of candidate biomarker TAC1 | 1 day
  Sensitivity of each candidate biomarker will be calculated by measuring the area under receiver operating characteristic curve generated from methylation index data.
Sensitivity of candidate biomarker HPP1 | 1 day
  Sensitivity of each candidate biomarker will be calculated by measuring the area under receiver operating characteristic curve generated from methylation index data.
Specificity of candidate biomarker p16 | 1 day
  Specificity of each candidate biomarker will be calculated by measuring the area under receiver operating characteristic curve generated from methylation index data.
Specificity of candidate biomarker NELL1 | 1 day
  Specificity of each candidate biomarker will be calculated by measuring the area under receiver operating characteristic curve generated from methylation index data.
Specificity of candidate biomarker AKAP12 | 1 day
  Specificity of each candidate biomarker will be calculated by measuring the area under receiver operating characteristic curve generated from methylation index data.
Specificity of candidate biomarker TAC1 | 1 day
  Specificity of each candidate biomarker will be calculated by measuring the area under receiver operating characteristic curve generated from methylation index data.
Specificity of candidate biomarker HPP1 | 1 day
  Specificity of each candidate biomarker will be calculated by measuring the area under receiver operating characteristic curve generated from methylation index data.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Meltzer, M.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland